CLINICAL TRIAL: NCT01330901
Title: UsTekinumab for the Treatment Of Patients With Active Ankylosing Spondylitis (TOPAS) - a 28-week, Prospective, Open-label, Proof-of-concept Study
Brief Title: Ustekinumab for the Treatment of Patients With Active Ankylosing Spondylitis
Acronym: TOPAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, J. Sieper, Prof. Dr., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOPAS
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ustekinumab (Experimental): Ustekinumab 90 mg subcutaneously at week 0, 4 and 16
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab 90 mg given subcutaneously at weeks 0, 4, and 16
  Other Names: Stelara

SUMMARY:
This study is aimed at investigation of efficacy and safety of ustekinumab (monoclonal antibody against interleukin 12 and 23) treatment in patients with active ankylosing spondylitis (AS) fulfilling the modified New York criteria who have had an inadequate response to standard therapy with non-steroidal anti-inflammatory drugs (NSAIDs) or do not tolerate or have a contraindication for NSAIDs.

DETAILED DESCRIPTION:
This study is a prospective, open-label, proof-of-concept clinical trial that will be conducted in a referral center for patients with AS in Berlin. Eligible patients will be treated with ustekinumab 90 mg given subcutaneously at weeks 0, 4, and 16. The entire study period accounts 28 weeks. Assessment of the primary outcome parameter will be performed at week 24. The patients will be closely monitored throughout the study on a total of 9 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥18 years.
2. Definite diagnosis of AS according to the modified New York criteria.
3. History of an inadequate response to ≥2 NSAIDs taken for at least 2 weeks each or NSAIDs intolerance/contraindication.
4. Active disease as defined by a BASDAI value of ≥4 at screening despite concomitant treatment with an NSAID or without NSAIDs in case of intolerance/contraindication.
5. Able and willing to give a written informed consent and comply with the requirements of the study protocol.
6. If female: either not of child-bearing potential (menopausal since 1 year or surgically sterile) or is willing and able to practice a reliable method of contraception.
7. If male: either not of child-bearing potential (surgically sterilized, e.g. vasectomy) or is willing and able to practice a reliable method of contraception.
8. If on NSAIDs: the dose must be stable for at least 2 weeks prior to baseline.
9. If on oral steroids: the dose must not exceed 10 mg (prednisolone equivalent) per day and must be stable for at least 4 weeks prior to baseline.
10. If on methotrexate: the dose must not exceed 25 mg per week and must be stable for at least 4 weeks prior to baseline, must be stable for 4 weeks prior to baseline.
11. If on analgesics: the dose must be stable for at least 2 weeks prior to baseline.

Exclusion Criteria:

1. The female subject is pregnant or lactating.
2. Patients with other chronic inflammatory articular disease or systemic autoimmune disease.
3. History of inadequate response to previous anti-tumor necrosis factor (TNF) α therapy.
4. Previous treatment with biologics other than TNF α blockers.
5. Treatment with any other investigational drug within 4 weeks of 5 half-life of the drug (whichever is longer) prior to baseline.
6. Treatments with disease modifying anti-rheumatic drugs (DMARDs) other than methotrexate within 4 weeks prior to screening (8 weeks for leflunomide or 4 weeks with a standard cholestyramine wash-out).
7. Treatment with intravenous, intramuscular or intraarticular/periarticular steroids within 4 weeks prior to screening.
8. Any active current infection, a history of recurrent clinically significant infection, infections requiring treatment with antibiotics within 4 weeks prior to baseline.
9. Current clinical signs and symptoms suggestive for tuberculosis.
10. Positive interferon gamma release assay (IGRA) test at screening and/or abnormal chest x-ray (performed at screening or within 3 months prior to screening) suggestive for past or present tuberculosis (positive x-ray). Patients with a positive IGRA test but negative chest x-ray and without clinical symptoms suggestive for tuberculosis may participate in the study after initiation of standard prophylactic antimycobacterial treatment.
11. Chronic infection with hepatitis B or C, history of human immunodeficiency virus infection.
12. Primary or secondary immunodeficiency.
13. Actual malignancies or history of malignancies with curative treatment within 5 years prior to screening, except successfully treated non-metastatic squamous-cell or basal-cell carcinoma or carcinoma in situ of the cervix.
14. Evidence of severe uncontrolled gastrointestinal, hepatic, renal, pulmonary, cardiovascular, nervous or endocrine disorders.
15. Any other conditions making the patient unsuitable in the opinion of the investigator for the participation in the current study.
16. Patients with a history of a severe psychiatric illness, which might interfere with the patient's ability to understand the requirements of the study and assessment.
17. Diagnosis of fibromyalgia.
18. Alcohol abuse or illegal drug consume in the last 12 months.
19. Vaccination with a live vaccine within 12 weeks prior to baseline.
20. Known hypersensitivity to any component of the study medication.
21. Clinically significant laboratory abnormalities
22. Patients who are institutionalised due to regulatory or juridical order.
23. Patients with contraindications for the magnetic resonance imaging (MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The Assessment of Spondyloarthritis International Society (ASAS)40 response | week 24
  The percentage of patients who achieved ASAS40 response defined as an improvement of ≥40% and ≥2 points in at least 3 out of four following domains (and no worsening in remaining domain):
  * Patient global
  * Pain
  * Function (as measured by the Bath Ankylosing Spondylitis Functional Index - BASFI)
  * Inflammation (mean of the Bath Ankylosing Spondylitis Disease Activity Index - BASDAI question 5 and 6)

SECONDARY OUTCOMES:
The Assessment of Spondyloarthritis International Society (ASAS)20 response at week 24 | Week 24
  The percentage of patients who achieved ASAS20 response defined as an improvement of ≥20% and ≥1 points in at least 3 out of four following domains (and no worsening of ≥20% and ≥1 points in remaining domain):
  * Patient global
  * Pain
  * Function (as measured by the Bath Ankylosing Spondylitis Functional Index - BASFI)
  * Inflammation (mean of the Bath Ankylosing Spondylitis Disease Activity Index - BASDAI question 5 and 6)
The Ankylosing Spondylitis Disease Activity Score (ASDAS) clinically important improvement | Week 24
  The percentage of patients who achieved the ASDAS clinically important improvement (≥1.1) at week 24
The Assessment of Spondyloarthritis International Society (ASAS) partial remission | Week 24
  The percentage of patients who achieved partial remission according to the ASAS definition at week 24
The Ankylosing Spondylitis Disease Activity Score (ASDAS) major improvement | Week 24
  The percentage of patients who achieved the ASDAS major improvement (≥2.0) at week 24
Number of participants with adverse events as a measure of safety and tolerability | Week 28
  Number of participants with adverse events as a measure of safety and tolerability up to week 28

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Rheumatology, Charité - Campus Benjamin Franklin, Berlin, Germany

REFERENCES:
- [Derived] Parthasarathy R, Santiago F, McCluskey P, Kaakoush NO, Tedla N, Wakefield D. The microbiome in HLA-B27-associated disease: implications for acute anterior uveitis and recommendations for future studies. Trends Microbiol. 2023 Feb;31(2):142-158. doi: 10.1016/j.tim.2022.08.008. Epub 2022 Sep 1. PMID 36058784
- [Derived] Poddubnyy D, Hermann KG, Callhoff J, Listing J, Sieper J. Ustekinumab for the treatment of patients with active ankylosing spondylitis: results of a 28-week, prospective, open-label, proof-of-concept study (TOPAS). Ann Rheum Dis. 2014 May;73(5):817-23. doi: 10.1136/annrheumdis-2013-204248. Epub 2014 Jan 3. PMID 24389297
- See also: Official web site of the study center — http://rheumatologie-berlin.de